CLINICAL TRIAL: NCT04141592
Title: Investigating Pathological Mechanisms in Non-alcoholic Fatty Liver Disease: Cross-sectional Comparative Study Between Patients and Healthy Controls
Brief Title: Investigating Pathological Mechanisms in Non-alcoholic Fatty Liver Disease
Status: Recruiting | Type: Observational
Sponsor: Queen Mary University of London (Other)
Collaborators: Homerton University Hospital NHS Foundation Trust (Other); Barts & The London NHS Trust (Other); King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 247449
Record Dates: First submitted 2019-10-23; First posted 2019-10-28 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — PBMCs, serum, plasma, liver tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Control: non-obese individuals without fatty liver disease
- Obese wihtout non-alcoholic steatohepatitis: Body mass index greater than 30 without liver histological evidence of non-alcoholic fatty liver disease
  Interventions: Procedure: Bariatric Surgery
- Obese Non-alcoholic steatohepatitis: Body mass index greater than 30 with liver histological evidence of non-alcoholic fatty liver disease
  Interventions: Procedure: Bariatric Surgery

INTERVENTIONS:
Procedure: Bariatric Surgery — Already clinically indicated surgical procedures
  Other Names: Upper GI surgery
  Groups: Obese Non-alcoholic steatohepatitis; Obese wihtout non-alcoholic steatohepatitis

SUMMARY:
To identify key characteristics of the tissue resident and peripherally circulating immune-phenotype in addition to blood markers, metabolic profile, faecal and oral microbiota in non-alcoholic fatty liver disease

DETAILED DESCRIPTION:
In this study, the investigators will collect tissue, blood, stool, urine and saliva samples at the same time in order to enable a comprehensive disease phenotyping and ability to compare immunological, microbiological and metabolic features in patients with varying stages of NAFLD and healthy controls. To date there are limited published data evaluating simultaneously-obtained samples from adipose, gut and liver tissue and peripheral blood in NAFLD. The majority of participants in this study will be recruited from the bariatric surgery services enabling multiple tissue samples to be collected at time of surgery with minimal additional risk to participants.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Confirmed non-alcoholic Fatty liver disease (diagnosed clinically, radiologically or histologically)
* If diabetic, Diagnosed with Type 2 Diabetes Mellitus

OR

• Healthy Control: no diagnosis of any liver condition including NAFLD

o NAFLD excluded by Fibroscan Controlled Attenuation Parameter (CAP) score of <222 dB/m

Exclusion Criteria:

* Unwilling or unable to give informed consent
* Type 1 Diabetes Mellitus
* Other form of liver disease (other than NAFLD)

  o Viral hepatitis, Auto-immune hepatitis, primary sclerosing cholangitis, primary biliary cholangitis, haemochromatosis, Sarcoidosis, cystic fibrosis, sickle cell disease
* Taking medication associated with liver dysfunction (except methotrexate)
* Auto-immune disease which in the investigator's opinion may confound immune profiling
* Concomitant immunosuppressive medications (except methotrexate, short course oral steroids or inhaled corticosteroids)
* Currently pregnant
* Any major organ transplant (excluding corneal or hair transplant)
* Regular alcohol intake greater than 14 units a week for female participants and 21 units a week for male participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be identified from outpatient clinics of Bariatric, Gastroenterology, and Hepatology services at Homerton and King College Hospitals in addition to Gastroenterology outpatients from the Barts Health NHS Trust. Healthy control participants will be identified from patients undergoing outpatient assessment, gastroscopy or surgery for other non-malignant gastrointestinal disorders at hospital sites.
Sampling Method: Probability Sample
Enrollment: 153 (Estimated)
Dates: Start 2019-03-05 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Impact of weight loss surgery upon Non-alcoholic steatohepatitis | Two years
  Proportion of patients developing resolution of NASH after weight loss surgery

SECONDARY OUTCOMES:
Impact of weight loss surgery upon Non-invasive measures of fibrosis | Six months
  Evaluation of changes in liver transient elastography post weight loss surgery

CONTACTS AND LOCATIONS:
Overall Officials: William Alazawi, MD Phd, Principal Investigator — Queen Mary University of London
Locations (1):
- Homerton University Hospital Foundation Trust, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/92/NCT04141592/Prot_000.pdf